CLINICAL TRIAL: NCT03813225
Title: Randomized Clinical Trial to Evaluate the Superiority on the Decrease the Consumption of Fentanyl the First 48 Hours of Bilateral Serratus Intercostal Plane Block in Myocardial Revascularization Surgery by Sternotomy.
Brief Title: Bilateral Serratus Intercostal Plane Block for Myocardial Revascularization (SERRINT)
Acronym: SERRINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Cardiovascular de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: fcv465
Record Dates: First submitted 2019-01-09; First posted 2019-01-23 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Pain, Postoperative; Pain Management; Analgesia, Patient-Controlled; Nerve Block
Keywords: Analgesia, patient- controlled, Block , Pain Postoperative
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Bites and Stings

STUDY DESIGN:
Intervention Model Description: Intervention: BILATERAL SERRATUS INTERCOSTAL- PLANE BLOCK plus usual multimodal analgesia
  Control:
  Usual multimodal analgesia
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant: The Patients will not know about intervention group they will be. Care Provider : The medical, nursing and pain clinical will not know the group to which the patient belongs Outcomes Assessor: during the analysis the staff will not know which group the patient belong
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Analgesia (No Intervention): These patients will receive the protocol multimodal analgesia patients receive on the Colombian Cardiovascular Foundation for handling an analgesic in cardiovascular surgery, this start in surgery with Lidocaine 0.5mcg/k. Dexamethasone 8mcg, Fentanyl Bolus: 7mcg/k . infusion of Fentanyl 4 mcg/k/h start after induction , go down to 2 Mcg/k/h during extracorporeal circulation , after extracorporeal circulation the infusion will be suspended of Fentanyl.
  and the postoperative analgesia will be 500mg of acetaminophen oral and Analgesia, patient controlled with Fentanyl 20mcg/bolus.
- Serrato intercostal plane Block (Experimental): These patients will receive the protocol multimodal analgesia patients receive on the Colombian Cardiovascular Foundation with Lidocaine 0.5mcg/k. Dexamethasone 8mcg, Fentanyl Bolus: 7mcg/k . infusion of Fentanyl 4 mcg/k/h start after induction , go down to 2 Mcg/k/h during extracorporeal circulation , after extracorporeal circulation the infusion will be suspended of Fentanyl.In this Arm the patient will give a bilateral serratus intercostal plane block, will be performed echo-guided puncture in the line anterior axillar with fifth costal arch, whit 21 ml of anesthetic mass, 20 ml of Levobupivacaine 0.375 and 1 mg (2mg) of dexamethasone. and the postoperative analgesia will be 500mg of acetaminophen oral and Analgesia, patient controlled with Fentanyl 20mcg/bolus
  Interventions: Other: Bilateral serratus Intercostal plane Block

INTERVENTIONS:
Other: Bilateral serratus Intercostal plane Block — Will be performed by echo guided one puncture in the fifth costal arch with anterior axilary line, where the tip of the needle will be guided until it reaches a point above the external intercostal muscle, below the anterior serratus above the costal arch where they will be administered 21 ml of anesthesic mass, (20 ml of levobupivacaine 0.375 and 1 mg (2mg) of dexamethasone.)
  Arms: Serrato intercostal plane Block

SUMMARY:
Two-parallel arm, double-blind, individually randomized controlled trial.

Primary endpoint:

Fentanyl consumption in the first 48 postoperative hours.

Secondary endpoints:

Pain at rest, Pain on movement, stay in ICU, Postoperative nausea and vomiting (PONV), sedation, Hemothorax, seizures, arrythmias

DETAILED DESCRIPTION:
Trial design: Two-parallel arm, double-blind, individually randomized controlled trial.

Primary endpoint:

Fentanyl consumption in the first 48 postoperative hours.

Secondary endpoints:

Pain at rest, Pain on movement, stay in ICU, Postoperative nausea and vomiting (PONV), sedation, Hemothorax, seizures, arrythmias

Inclusion criteria:

* Patient between 18 years to 80 years.
* Patient to myocardial revascularization by sternotomy

Exclusion criteria:

* Patitient for combined surgery ( myocardial revascularization by sternotomy plus valve or maze)
* Emergency surgery
* Ejecction Fraction less than 35%
* Allergy to the local anesthesic.
* Allergy to opioids
* Patient in who will be technically impossible the application of the blockade

Trial treatment:

Intervention: These patients will receive the protocol multimodal analgesia patients receive on the Colombian Cardiovascular Foundation with Lidocaine 0.5mcg/k. Dexamethasone 8mcg, Fentanyl Bolus: 7mcg/k . infusion of Fentanyl 4 mcg/k/h start after induction , go down to 2 Mcg/k/h during extracorporeal circulation , after extracorporeal circulation the infusion will be suspended of Fentanyl.In this Arm the patient will give a bilateral serratus intercostal plane block, will be performed echo-guided puncture in the line anterior axillar with fifth costal arch, whit 21 ml of anesthetic mass, 20 ml of Levobupivacaine 0.375 and 1 ml (2mg) of dexamethasone. and the postoperative analgesia will be 500mg of acetaminophen oral and Analgesia, patient controlled with Fentanyl 20mcg/bolus

Control:

These patients will receive the protocol multimodal analgesia patients receive on the Colombian Cardiovascular Foundation with Lidocaine 0.5mcg/k. Dexamethasone 8mcg, Fentanyl Bolus: 7mcg/k . infusion of Fentanyl 4 mcg/k/h start after induction , go down to 2 Mcg/k/h during extracorporeal circulation , after extracorporeal circulation the infusion will be suspended of Fentanyl.. and the postoperative analgesia will be 500mg of acetaminophen oral and Analgesia, patient controlled with Fentanyl 20mcg/bolus

Expected sample size, enrollment and expected number of centers:

Sample size = 44 Recruitment start date: 15 january of 2019 Recruitment end date: 15 July of 2019

Follow-up end date:

Number of centers: 1

Statistical considerations:

* Intention to treat analysis
* The primary outcomes will be analyzed using

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 years to 80 years
* Patient to myocardial revascularization by sternotomy

Exclusion Criteria:

* Patient for combined surgery ( myocardial revascularization by sternotomy plus valve or maze)
* Emergency surgery
* Ejection Fraction less than 35%
* Allergy to the local anesthesics.
* Allergy to opioids
* Patient in who will be technically impossible the application of the blockade

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Fentanyl Consume | 48 hours
  Microgrames of Fentanyl that patient consume during the first 48 hours in the postoperative

SECONDARY OUTCOMES:
Pain In Rest and in motion | 48 hours
  It will be valued the pain at rest and in motion, by means of the verbal analog scale for pain, where zero is the absence of pain and 10 is the worst pain that has had on the lives, the pain is measured from the time of extubation what we will call zero hour, and every four hours per 48 hours.
Nausea and vomiting | 48 hours.
  Presence of nausea and vomiting during the first 48 hours postoperative.
Sedation | 48 hours.
  Assessment of sedation in the first 48 hours postoperative with the Ramsay scale .The Ramsay scale , Is a subjective scale to assess the degree of sedation of patients, values 6 levels, from 1 where the patient is anxious and agitated ,2 Awake, coperador, focused and quiet. 3. Slept with response to orders. 4. Sleepy with brief answers to the Light. 5 is patient Slept with an answer only to the pain and 6 where the patient is deep asleep without response to stimuli.
hemothorax | 24 hours
  presence of hemothorax secundary to blockage
seizures | 1 hour after block
  presence of seizure after to blockage
Arrhythmias | 1 hour after block
  presence of Arrhythmias after of blockage

CONTACTS AND LOCATIONS:
Overall Officials: luz Pacheco, Esp, Principal Investigator — Fundacion Cardiovascular
Locations (1):
- Luz Jenny Pacheco, Floridablanca, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No